CLINICAL TRIAL: NCT07365423
Title: Terbinafine for Biochemically Recurrent Prostate Cancer (TerbinaPro) - A Phase II Drug-repurposing Study
Brief Title: Terbinafine for Biochemically Recurrent Prostate Cancer (TerbinaPro)
Acronym: TerbinaPro
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCI 001
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Prostate Cancer
Keywords: recurrent prostate cancer; Terbinafine; phase II; drug-repurposing Study
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Terbinafine

STUDY DESIGN:
Intervention Model Description: Open label, two-stage design with three dose levels Patients with biochemically recurrent Prostate Cancer (PCa) after exhaustion of local treatment options with curative intent with non-castrate levels of testosterone will be randomized to treatment with Terbinafine either at the licensed dose of 250 mg daily or an escalated dose of 500 mg or 1000 mg daily for up to 12 cycles, consisting of 28 days each. In stage I, all three dose levels will be opened and enrolled in parallel. Additional patients will be enrolled in stage II, at a selected dose level, based on the results obtained in Stage I.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1 (Experimental): Patients will be randomized in a 1:1:1 ratio for a total of 9 patients per dose level to either the standard dose (250mg) or an escalated dose (500mg or 1000mg).Treatment duration: up to 12 cycles of 28 days
  Interventions: Drug: Terbinafine
- Stage 2 (Experimental): Additional patients will be enrolled in stage II, at a selected dose level, based on the results obtained in Stage I.
  Treatment duration: up to 12 cycles of 28 days
  Interventions: Drug: Terbinafine

INTERVENTIONS:
Drug: Terbinafine — Drug: Terbinafine

SUMMARY:
TerbinaPro is a phase II drug-repurposing study evaluating oral Terbinafine in patients with biochemical recurrence of prostate cancer after prior local treatment with curative intent. When local salvage strategies have been exhausted, recurrence usually reflects micro-metastatic disease without clearly visible metastases on imaging. Standard therapy with androgen deprivation or androgen-receptor pathway inhibitors can effectively control disease but is associated with substantial side effects and negative impact on quality of life. Terbinafine is a long-licensed, generic antifungal drug that inhibits squalene epoxidase (SQLE), an enzyme that may play a role in prostate cancer progression. Preclinical and limited clinical data suggest potential anti-cancer activity.

DETAILED DESCRIPTION:
About 20-50% of patients with prostate cancer will develop biochemical recurrence within 10 years after local treatment with initial curative intent. After exhaustion of local salvage strategies such as radiotherapy to the prostate bed, biochemical recurrence usually indicates micro metastatic locoregional or distant disease, mostly no longer amenable to curative strategies. Evidence on how to treat these patients without clearly visible metastatic disease on imaging is very limited. Eventually, patients will be started on androgen deprivation therapy and/or androgen-receptor pathway inhibitors. These treatments however have well-known side effects and negative impact on quality of life such as causing hot flushes, reduction of bone and muscle mass and affecting sexual function and psychological wellbeing. Many patients therefore have an interest to postpone initiation of androgen deprivation and new treatment options are needed. Terbinafine is a long-licensed and generic anti-fungal drug used to treat fungal infections of nails and skin with a very favorable side-effect profile. Its mode of action is inhibition of the fungal enzyme squalene epoxidase (SQLE) which results in accumulation of squalene and consecutive fungal cell death. SQLE is also present in mammalian cells and a growing amount of preclinical and limited clinical study data suggests that SQLE may play a role in development and progression of different cancer types. In prostate cancer, overexpression of SQLE has been documented and shown to be associated with adverse outcomes. Tissue culture and xenograft models show inhibition of prostate cancer cells by Terbinafine, including models resistant to androgen-receptor pathway inhibitors. Limited clinical and retrospective population-based data also suggest activity of Terbinafine in patients with prostate cancer. However, so far, the drug has not been tested systematically in prostate cancer patients and based on our knowledge, no such trials are currently ongoing. TerbinaPro is a drug repurposing phase II study to assess activity of Terbinafine in biochemical recurrence of prostate cancer.

The primary objective of the trial is to demonstrate efficacy of Terbinafine in biochemically recurrent prostate cancer. Secondary objectives are exploration of an active oncological dose and safety of treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients after definitive treatment for localized prostate cancer and exhaustion of standard curative options (i.e. after prostatectomy and adjuvant /salvage radiotherapy; definite radiotherapy, brachytherapy; additional previous Stereotactic Body Radiation Therapy (SBRT) to treat visible oligometastatic disease also allowed as long as confirmed Prostate-specific antigen (PSA) progression is present after SBRT)
* Non-castrate levels of testosterone (≥ 5 nmol/l; previous androgen deprivation therapy (ADT) allowed as long as testosterone levels have recovered before study entry)
* No evidence of distant metastatic disease on conventional imaging (Computed Tomography (CT) and bone scan) or Prostate-Specific Membrane Antigen (PSMA) Positron Emission Tomography (PET) CT.
* Patients with PSMA positive lymph nodes on PSMA PET CT can still be included if the short axis of the largest lymph node is < 20 mm for lymph nodes below aortic bifurcation or < 10 mm above the aortic bifurcation.
* PSA of ≥1 ng/ml after radical prostatectomy or ≥2 ng/ml above the nadir (with recovered testosterone) after primary radiotherapy; confirmation of rising PSA in at least a second measurement at least 2 weeks apart
* Patient declining start of ADT and /or an androgen receptor pathway inhibitor (ARPI) and/or judged as not in need of immediate ADT/ARPI start by treating physician

Key Exclusion Criteria:

* Pre-existing known chronic or acute liver disease
* Known history of systemic lupus erythematosus or any form of lupus (including cutaneous, drug-induced, or lupus nephritis)
* Pure neuroendocrine/small-cell histologic variant of prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Prostate specific antigen Progression-free rate (PSA-PFR) | From the date of treatment start until 12 weeks after treatment start
  The primary endpoint is PSA-PFR at week 12 from start of treatment with Terbinafine. To calculate PSA-PFR at week 12, the Kaplan-Meier estimator of time to PSA progression will be evaluated at 13 weeks after treatment start, to allow 1 week delay in the assessment at 12 weeks.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of treatment start until the date of progression or death from any cause, assessed up to 1 year after end of treatment.
  PFS will be calculated from treatment start until one of the following events, whichever occurs first:
  * Death from any cause
  * Presence of unequivocal radiographic progression as assessed by the local investigator
  * Presence of PSA progression
  * Presence of clinical/symptomatic progression Patients without an event will be censored at the date of the last available assessment showing no event before the start of the subsequent treatment, if any.
Prostate-specific antigen (PSA) response (30%, 50%, 90% and best) | From the date of treatment start until the end of treatment, estimated up to 336 days after treatment start.
  * 30% PSA response is defined as a decrease in PSA level of at least 30% (compared to baseline PSA).
  * 50% PSA response is defined as a decrease in PSA level of at least 50% (compared to baseline PSA).
  * 90% PSA response is defined as a decrease in PSA level of at least 90% (compared to baseline PSA).
  Best PSA response is defined as the percentage of change in PSA from baseline to the maximum decline in PSA at any point under treatment. If there is a steady increase after baseline, the best response is defined as the percentage of change in PSA from baseline to the minimum increase in PSA at any point under treatment. Baseline is defined as the latest recorded PSA measurement prior to the first dose of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Fischer, PD MD, Study Chair — HOCH Health Ostschweiz; Richard Cathomas, Prof, Study Director — Cantonal Hospital Graubünden
Locations (12):
- Switzerland (12):
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - EOC - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Kantonsspital Graubünden, Chur
  - Spital Thurgau AG, Frauenfeld
  - Hôpitaux Universitaires Genève HUG, Geneva
  - Luzerner Kantonsspital, Lucerne
  - TBZO Tumor- und BrustZentrum Ostschweiz - Rapperswil, Rapperswil
  - HOCH Health Ostschweiz - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Universitätsspital Zürich USZ, Zurich